CLINICAL TRIAL: NCT00501475
Title: NAC in Preventing CIN in CRF Patients Who Need Enhanced CT Scan in ED
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06-2006-084
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Chronic Renal Failure
Keywords: N-acetylcysteine; nephropathy; bicarbonate
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: NAC Bicarbonate

SUMMARY:
The purpose of this study is to evaluate the effect of NAC or sodium bicarbonate in preventing the aggravation of renal function in chronic renal failure when enhanced computed tomography scan is checked in emergency room.

DETAILED DESCRIPTION:
CIN is frequent in CRF patients. However most studies about CIN has been focusing on elective PCI patients. There is no study that the NAC nor sodium bicarbonate would help in preventing CIN in CRF patients who need enhanced CT scan in ED.

Our intention was to investigate the effect of NAC or sodium bicarbonate in preventing the aggravation of renal function in chronic renal failure when enhanced computed tomography scan is checked in emergency room.

ELIGIBILITY:
Inclusion Criteria:

* CRF patients who need enhanced CT scan

Exclusion Criteria:

* less than 15 years old
* hypersensitivity to NAC
* on dialysis
* no consent from patient or next of kin

Min Age: 15 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-03; Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
the rate of CIN | 3 days after CT scan

SECONDARY OUTCOMES:
mortality | 30 days after CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Kyuseok Kim, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul, 28 Yongon-dong, Chongro-gudo
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeongi-do